CLINICAL TRIAL: NCT06500663
Title: Studying Thyroid Function of Haemodialysis Patients in Upper Egypt (Two Centers Study).
Status: Not yet recruiting | Type: Observational
Sponsor: Sahar Ezeldeen Hussein Ali (Other)
Collaborators: Assiut University (Other)
Responsible Party: Sponsor-Investigator, Sahar Ezeldeen Hussein Ali, Assuit, Assiut University
Organization: Assiut University (Other)
Other Study IDs: DR.sahar protocol; faculty (Other: of medicine Assuit university)
Record Dates: First submitted 2024-07-08; First posted 2024-07-15 (Actual); Last update posted 2024-07-15 (Actual); Status verified 2024-07

CONDITIONS: Haemodialysis Patients
MeSH Terms: interventions — Dialysis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- 1: patients on haemodialysis themselves and their hospital records including the participant's information (name, age, sex, admission date, clinical procedures, medications administered…etc).
  Interventions: Other: haemodialysis

INTERVENTIONS:
Other: haemodialysis — haemodialysis effect on thyroid function

SUMMARY:
1. The study aims to investigate the prevalence of thyroid dysfunction in haemodialysis patients and study the association of thyroid hormone concentration with health status of those patients
2. Study the effects of frequent haemodialysis on thyroid function

DETAILED DESCRIPTION:
2.1 Background (Research Question, Available Data from the literature, Current strategy for dealing with the problem, Rationale of the research that paves the way to the aim(s) of the work). (200-250 words max.) The study of thyroid function in hemodialysis patients is a critical area of research due to the complex interplay between renal failure and thyroid pathology. Chronic kidney disease (CKD) and end-stage renal disease (ESRD) have been associated with various thyroid abnormalities, including hypothyroidism and low triiodothyronine (T3) syndrome (1). These conditions can significantly impact the morbidity and mortality of patients undergoing hemodialysis (2).

In hemodialysis patients, the prevalence of thyroid dysfunction is higher compared to the general population(3). This is partly due to the altered metabolism and clearance of thyroid hormones and the impact of uremic toxins on thyroid function (4). Moreover, thyroid hormones play a crucial role in cardiovascular health, which is of particular concern in hemodialysis patients who are already at an increased risk for cardiovascular events (5).

Recent studies have shown that even subclinical hypothyroidism, where patients have an elevated thyroid-stimulating hormone (TSH) level but normal thyroxine (T4) levels, can be associated with adverse outcomes in hemodialysis patients (6). This condition may contribute to an increased risk of cardiovascular disease and mortality (7).

The assessment of thyroid function in hemodialysis patients typically involves measuring serum levels of TSH, free T4, and T3 (8). However, interpreting these levels can be challenging due to the effects of medications, nutritional status, and non-thyroidal illness on the thyroid axis (9). It is also important to consider the impact of hemodilution on thyroid function tests, as it can lead to misinterpretation of the results (10).

Management of thyroid dysfunction in hemodialysis patients requires careful consideration. While thyroid hormone replacement therapy is commonly used to treat hypothyroidism, the optimal target levels of TSH and T4 in this population are still under investigation (11). Additionally, the benefits of treating subclinical hypothyroidism in hemodialysis patients remain uncertain (12).

In the context of Egypt, the prevalence of thyroid dysfunction among hemodialysis patients mirrors global trends. A study conducted in a South Indian cohort, which may have parallels in Egypt due to similar dietary and environmental factors, found a high prevalence of subclinical hypothyroidism in hemodialysis patients(13). This suggests that thyroid screening and management should be an integral part of care for hemodialysis patients in Egypt as well.

Egypt's healthcare system has been making strides in improving the management of chronic diseases, including CKD and its complications. With a growing focus on preventive care and early intervention, the management of thyroid dysfunction in hemodialysis patients is likely to receive more attention in the coming years (14).

In Upper Egypt, research has been conducted to investigate the prevalence and nature of thyroid abnormalities among hemodialysis patients. A cross-sectional observational report enrolled 160 subjects at Al-Hussein Hospital, Al-Azhar University, and the National Institute of Nephrology and Urology, revealing significant correlations between thyroid hormones and various clinical parameters (15). Another study assessed thyroid hormone levels in 200 patients with chronic renal failure undergoing maintenance hemodialysis, finding a high prevalence of thyroid hormone dysfunction even in clinically euthyroid patients(16).

In conclusion, the study of thyroid function in hemodialysis patients is essential for optimizing patient outcomes. With ongoing research and improved clinical practices, the management of thyroid dysfunction in this vulnerable population can be enhanced. As Egypt continues to develop its healthcare infrastructure, it is poised to make significant contributions to this field of study (17).

ELIGIBILITY:
Inclusion Criteria:

1. Patients who have been on hemodialysis for at least 6 months.
2. Patients aged between 18 and 75 years
3. Patients without overt hyper/hypothyroidism or thyroid hormone supplementation (for examining endogenous thyroid function).

Exclusion Criteria:

- 4. Patients with a history of thyroid disease or thyroid surgery. 5. Patients currently on medications known to affect thyroid function (e.g., amiodarone, lithium).

6. Pregnant or breastfeeding women. 7. Patients with other serious illnesses (e.g., cancer, severe heart disease) that could affect thyroid function or the ability to participate in the study 8. Patients receiving thyroid hormone supplementation

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: based on determining the main outcome variable, The estimated minimum required sample size is 160 patients. The sample size was calculated using Epi-info version 7 software, based on the following assumptions: Main outcome variable is which is to investigate the prevalence of thyroid disfunction in haemodialysis patients and the association of thyroid hormone concentration with health status of those patients Based on previous studies (Lo et al., 2017) the prevalence of thyroid disfunction in haemodialysis patients was 21.8% , and based on the percentage confidence limits of 4% and a Confidence level =80% .
Sampling Method: Probability Sample
Enrollment: 160 (Estimated)
Dates: Start 2024-08-01 (Estimated); Primary Completion 2025-12-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
1. Prevalence of Hypothyroidism: The primary outcome measure could be the prevalence of hypothyroidism in patients with end-stage renal disease (ESRD) undergoing frequent hemodialysis | 1 year
  2. Changes in Thyroid Hormone Levels: Another primary outcome measure could be the changes in serum TSH, free thyroxine (FT4), and free triiodothyronine (FT3) concentrations in patients undergoing frequent hemodialysis.

SECONDARY OUTCOMES:
1. Correlation of TSH Concentrations with Age: A secondary outcome measure could be the correlation of TSH concentrations with age. | 1 year
  2. Association of Thyroid Hormone Levels with Health Status: the association of circulating thyroid hormone levels with parameters of self-reported health status, and physical and cognitive performance.
  3. Effects of Increased Dialysis Frequency on Thyroid Indices: The effects of increased dialysis frequency on thyroid indices in patients receiving haemodialysis without overt hyper/hypothyroidism or thyroid hormone treatment.

IPD SHARING:
Plan to Share IPD: Undecided
1. The study aims to investigate the prevalence of thyroid dysfunction in haemodialysis patients and study the association of thyroid hormone concentration with health status of those patients
  2. Study the effects of frequent haemodialysis on thyroid function..

REFERENCES:
- [Background] Lo JC, Chertow GM, Go AS, Hsu CY. Increased prevalence of subclinical and clinical hypothyroidism in persons with chronic kidney disease. Kidney Int. 2005 Mar;67(3):1047-52. doi: 10.1111/j.1523-1755.2005.00169.x. PMID 15698444
- [Background] Kaptein EM, Quion-Verde H, Chooljian CJ, Tang WW, Friedman PE, Rodriquez HJ, Massry SG. The thyroid in end-stage renal disease. Medicine (Baltimore). 1988 May;67(3):187-97. doi: 10.1097/00005792-198805000-00005. PMID 3259281
- [Background] Lim VS. Thyroid function in patients with chronic renal failure. Am J Kidney Dis. 2001 Oct;38(4 Suppl 1):S80-4. doi: 10.1053/ajkd.2001.27410. PMID 11576928
- [Background] Schultheiss UT, Steinbrenner I, Nauck M, Schneider MP, Kotsis F, Baid-Agrawal S, Schaeffner E, Eckardt KU, Kottgen A, Sekula P; GCKD investigators. Thyroid function, renal events and mortality in chronic kidney disease patients: the German Chronic Kidney Disease study. Clin Kidney J. 2020 Jun 4;14(3):959-968. doi: 10.1093/ckj/sfaa052. eCollection 2021 Mar. PMID 34349984
- [Background] Sanai T, Okamura K, Onoue T, Ono T, Motomura K, Miyazono M, Shimamatsu K. Hemodilution Impacts Assessment of Thyroid Status before and after Hemodialysis in Patients with End-Stage Renal Disease. Am J Nephrol. 2021 Feb 1;51(12):988-994. doi: 10.1159/000512968. Online ahead of print. PMID 33524972
- [Background] Rhee CM, You AS, Nguyen DV, Brunelli SM, Budoff MJ, Streja E, Nakata T, Kovesdy CP, Brent GA, Kalantar-Zadeh K. Thyroid Status and Mortality in a Prospective Hemodialysis Cohort. J Clin Endocrinol Metab. 2017 May 1;102(5):1568-1577. doi: 10.1210/jc.2016-3616. PMID 28324018